CLINICAL TRIAL: NCT01975857
Title: Evaluating a Novel Sleep-focused Mind-body Rehabilitative Program for Veterans With mTBI and Other "Polytrauma" Symptoms: An Randomized Controlled Trial (RCT) Study
Brief Title: Mind-Body Rehabilitative Program for Veterans With mTBI (Mild Traumatic Brain Injury)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: VA Salt Lake City Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Yoshio Nakamura, Research Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00061854
Record Dates: First submitted 2013-07-08; First posted 2013-11-05 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Sleep Disturbance; Traumatic Brain Injury
Keywords: mild traumatic brain injury; sleep; mind body intervention; mind body bridging
MeSH Terms: conditions — Parasomnias; Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mind-Body Bridging Program (Experimental): The Mind-Body Bridging Program (MBBP) is an awareness training program (ATP) to help individuals improve their health condition and attain a state of well-being. Bridging is the primary technique that facilitates the healing process, by bringing one back to the present moment to experience thoughts, emotions and physical sensations. Bridging aims to reduce the impact of negative thought patterns that contribute to stress in the body.
  Interventions: Behavioral: Mind-Body Bridging Program
- Supportive Education (Active Comparator): Supportive Education program will provide educational lectures on disability, sleep hygiene, and current research on depression and non-directive, supportive discussions about these topics.
  Interventions: Behavioral: Supportive Education

INTERVENTIONS:
Behavioral: Mind-Body Bridging Program — Bridging aims to reduce the impact of negative thought patterns that contribute to stress in the body.
  Other Names: MBB
  Arms: Mind-Body Bridging Program
Behavioral: Supportive Education — This intervention will provide educational lectures on disability, sleep hygiene, and current research on depression and nondirective, supportive discussions about these topics.
  Other Names: SED
  Arms: Supportive Education

SUMMARY:
The broad aim of the proposed study is to evaluate the comprehensive benefit of a novel mind-body therapeutic intervention, Mind-Body Bridging (MBB), in Veterans who suffer from mTBI and sleep disturbance co-morbid with PTSD and/or pain at the VA Salt Lake City Health Care System (VASLCHCS). Evidence for comprehensive benefit includes, but is not limited to, the average difference in outcomes between MBB and an active control, sleep education (SED), both integrated with the usual care for mTBI Veterans. The long-term goal of the proposed project is to introduce, implement and establish mind-body intervention programs as a behavioral health intervention modality that would serve as a generally sustainable health care intervention program before, during, and after deployment for military personnel.

DETAILED DESCRIPTION:
Traumatic brain injury represents a dynamic spectrum of physiologic and cognitive dysfunction that exerts effects at multiple levels of human health. Mild traumatic brain injury (mTBI) is a multi-factorial illness that is an increasingly serious public health issue for military and civilian personnel. The assessment of neurocognitive deficits in mTBI has been suggested to be less conclusive, presumably because of the predominating influence of PTSD and other co-morbid factors. Recent research suggests that psychological factors play a substantial role in TBI-related impairments in self-reported health and cognition function. Furthermore, research has shown that TBI is rarely an isolated finding in military combat settings and that persistent post-concussive symptoms are commonly associated with post-traumatic stress disorder and chronic pain, a constellation of findings that has been termed the "polytrauma clinical triad". Indeed, significant numbers of returning Veterans of Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) display the polytrauma clinical triad (PCT) of pain, posttraumatic stress disorder (PTSD), and traumatic brain injury. The proposed project will: 1) elucidate best practices for treating mTBI with co-occurring symptoms (pain, sleep disturbance, PTSD) encompassing cognitive, emotional, and psychological functioning; and 2) address psychosocial aspects of managing pain and co-morbidities associated with mTBI through integrative and complementary and alternative approaches.

ELIGIBILITY:
Inclusion Criteria:

* Veteran from OEF/OIF
* has been diagnosed with mTBI
* has current sleep disturbance as indicated by a score of 35 or greater on the MOS-Sleep Scale (MOS-SS)

Exclusion Criteria:

* serious psychiatric comorbidity
* active intense suicidal intent
* inpatient admission to psychiatric ward in the last 3 month
* the presence of co-occurring progressive/advanced neurodegenerative disease
* terminally ill
* unstable chronic medical conditions
* untreated sleep apnea
* presence of substance dependence disorder
* narcolepsy
* frequent nocturia
* delayed sleep phase syndrome
* advanced sleep phase syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Change in self-reported measures of sleep using Medical Outcomes Study -Sleep Scale, from baseline (Pre) to 6 months follow-up | Pre (within one month before Intervention week 1), Intervention week 1, Intervention week 2, Intervention week 3, Post (one week after Intervention week 3), 3 month Follow-up, 6 month Follow-up
  The Medical Outcomes Study Sleep Scale (MOS-SS) provides an index of sleep problems and incorporates six sleep scale scores: 1) sleep disturbance, 2) sleep adequacy, 3) daytime somnolence, 4) snoring, 5) waking up short of breath with a headache, and 6) quantity of sleep. The MOS-SS is similar to the Pittsburgh Sleep Quality Index (PSQI) developed at the same time, which includes more questions about sleep disturbance with seven more items overall. The 1-week assessment is adapted from the normal 4-week retrospective assessment.
Change in latency to sleep onset using the Sleep Diary, from baseline (Pre) to 6 months follow-up. | Pre (within one month before Intervention week 1), Intervention week 2, Post (one week after Intervention week 3), 3 month Follow-up, 6 month Follow-up
  The Sleep Diary is a commonly used self-reported sleep assessment measure. Participants will be asked to complete a sleep diary for seven days. In the sleep diary, participants will record different daily events and activities (e.g., the number of times they wake up during the night, whether they have been drinking caffeinated beverages, or exercising). Sleep-related entries include recording when they go to bed, when they think they fell asleep, duration of sleep, and naps during the day.
Change in self-reported mTBI symptoms using the Neurobehavioral Symptom Inventory (NSI), from baseline (Pre) to 6 months follow-up. | Pre (within one month before Intervention week 1), Post (one week after Intervention week 3), 3 month Follow-up, 6 month Follow-up
  The NSI is a self-report measure of post-concussive symptoms comprising 22-items. Participants rate the degree of symptom severity on a five-point scale ranging from 0 (none) to 4 (very severe) over the past 2 weeks. The NSI total score is the sum of severity ratings of the 22 symptoms, and ranges from 0 to 88. The NSI reflects a 9 symptom cluster model, which can be validly reduced to 3 clusters, namely, cognitive, affective, and somatic/sensory symptoms.
Change in self-reported Quality of Life using the Medical Outcomes Study (MOS) Short Form-36 (SF-36) for Veterans (MOS SF-36V), from baseline (Pre) to 6 months follow-up. | Pre (within one month before Intervention week 1), Post (one week after Intervention week 3), 3 month Follow-up, 6 month Follow-up
  The MOS SF-36V is a well-established standard measure of quality of life (QOL) scale, to assess mental and physical health as well as functional status, adapted for Veterans. The MOS SF-36V consists of the same eight sections as the civilian version, MOS SF-36. Higher scores indicate better quality of life. The instrument provides a global score, as well as the following subscale scores: functional capacity, physical aspects, pain, general health condition, vitality, social aspects and emotional aspects, and mental health.
Change in duration of sleep using the Sleep Diary, from baseline (Pre) to 6 months follow-up. | Pre (within one month before Intervention week 1), Intervention week 2, Post (one week after Intervention week 3), 3 month Follow-up, 6 month Follow-up
  The Sleep Diary is a commonly used self-reported sleep assessment measure. Participants will be asked to complete a sleep diary for seven days. In the sleep diary, participants will record different daily events and activities (e.g., the number of times they wake up during the night, whether they have been drinking caffeinated beverages, or exercising). Sleep-related entries include recording when they go to bed, when they think they fell asleep, duration of sleep, and naps during the day.
Change in number of awakenings using the Sleep Diary, from baseline (Pre) to 6 months follow-up. | Pre (within one month before Intervention week 1), Intervention week 2, Post (one week after Intervention week 3), 3 month Follow-up, 6 month Follow-up
  The Sleep Diary is a commonly used self-reported sleep assessment measure. Participants will be asked to complete a sleep diary for seven days. In the sleep diary, participants will record different daily events and activities (e.g., the number of times they wake up during the night, whether they have been drinking caffeinated beverages, or exercising). Sleep-related entries include recording when they go to bed, when they think they fell asleep, duration of sleep, and naps during the day.
Change in physical activity during sleep for assessment of sleep quality using a heart rate and motion detection device, from baseline (Pre) to 3 months follow-up | Pre (within one month before Intervention week 1), Post (one week after Intervention week 3), 3 month Follow-up
  The non-invasive heart rate and motion detection device will be used to quantify physical activity during sleep for assessment of sleep quality as a measure of sleep disturbance. Each participant will be asked to wear the device for 2 consecutive days of home assessment.
Change in heart rate variability for assessment of sleep quality using a heart rate and motion detection device, from baseline (Pre) to 3 months follow-up | Pre (within one month before Intervention week 1), Post (one week after Intervention week 3), 3 month Follow-up
  The non-invasive heart rate and motion detection device will be used to quantify heart rate variability for assessment of sleep quality as a measure of sleep disturbance. Each participant will be asked to wear the device for 2 consecutive days of home assessment.

SECONDARY OUTCOMES:
Change in self-reported PTSD using the PTSD Checklist - Military Version (PCL-M), from baseline (Pre) to 6 months follow-up. | Pre (within one month before Intervention week 1), Post (one week after Intervention week 3), 3 month Follow-up, 6 month Follow-up
  The PCL-M is a well-validated 17-item self-report measure to assess PTSD severity among military personnel; both male and female, to assess military-related PTSD. Reliability evidence is very good. Items are based on DSM criteria (DSM-IV criteria for the latest version) and are rated on a 5-point Likert-type scale that allows the derivation of a quantifiable total score.
Change in self-reported pain symptoms using the Brief Pain Inventory (BPI), from baseline (Pre) to 6 months follow-up. | Pre (within one month before Intervention week 1), Post (one week after Intervention week 3), 3 month Follow-up, 6 month Follow-up
  The BPI is one of the most widely used instruments for assessing clinical pain. Patients rate their current pain intensity and also pain in the last 24 hours at its worst, least, and average by using a numeric scale of 0 (no pain) to 10 (pain as bad as you can imagine). Patients also rate the extent to which their pain interferes with 7 quality of life domains identifying how they feel and their functionality, e.g., general activity, walking, mood, sleep, work, relations with other persons, and enjoyment of life.
Change in self-reported depression symptoms using the Center for Epidemiologic Studies Depression Scale (CES-D), from baseline (Pre) to 6 months follow-up. | Pre (within one month before Intervention week 1), Post (one week after Intervention week 3), 3 month Follow-up, 6 month Follow-up
  The CES-D is one of the most common validated screening tests for helping an individual to determine their depression quotient. The 20-item test measures depressive feelings and behaviors during the past week.
Change in self-reported resilience using the Connor-Davidson Resilience Scale (CD-RISC), from baseline (Pre) to 6 months follow-up. | Pre (within one month before Intervention week 1), Post (one week after Intervention week 3), 3 month Follow-up, 6 month Follow-up
  One of the few well-validated measures of resilience is the Connor-Davidson Resilience Scale (CD-RISC), comprising 25 items.
Change in self-reported perceived stress symptoms using the Perceived Stress Scale (PSS), from baseline (Pre) to 6 months follow-up. | Pre (within one month before Intervention week 1), InterventionWeek1, InterventionWeek2, InterventionWeek3, Post (one week after Intervention week 3), 3 month Follow-up, 6 month Follow-up
  The PSS measures the degree to which participants consider situations to be stressful, based on the extent to which they perceive their lives to be unpredictable, uncontrollable, or overloaded. It measures the amount of stress in one's life rather than response to a specific stressor.
Change in self-reported self-compassion using the Self-Compassion Scale (SCS), from baseline (Pre) to 6 months follow-up. | Pre (within one month before Intervention week 1), Post (one week after Intervention week 3), 3 month Follow-up, 6 month Follow-up
  The SCS comprises 26 items and is used to measure self-compassion, an emotionally positive self-attitude that should protect against the negative consequences of self-judgment, isolation, and rumination (such as depression). Self-compassion seems to entail three main components: 1) self-kindness, being kind and understanding toward oneself in instances of pain or failure rather than being harshly self-critical, 2) common humanity, perceiving one's experiences as part of the larger human experience rather than seeing them as separating and isolating, and 3) mindfulness, holding painful thoughts and feelings in balanced awareness rather than over-identifying with them. Thus, SCS may be used to assess the potential benefits induced by mindfulness based interventions, which may be strongly related to the construct of self-compassion.
Change in self-reported mindfulness using the Five Facet Mindfulness Questionnaire (FF-MQ), from baseline (Pre) to 6 months follow-up. | Pre (within one month before Intervention week 1), InterventionWeek1, InterventionWeek2, InterventionWeek3, Post (one week after Intervention week 3), 3 month Follow-up, 6 month Follow-up
  The FF-MQ includes 39 items and assesses five distinct, interpretable facets of mindfulness, including: 1) observing, 2) describing, 3) acting with awareness, 4) non-judging of inner experience, and 5) non-reactivity to inner experience.
Change in self-reported well-being using the Well-Being Index (WBI), from baseline (Pre) to 6 months follow-up. | Pre (within one month before Intervention week 1), InterventionWeek1, InterventionWeek2, InterventionWeek3, Post (one week after Intervention week 3), 3 month Follow-up, 6 month Follow-up
  The WBI is a five item scale evaluating both positive and negative aspects of emotional functioning, developed and validated by the World Health Organization Collaborating Centre in Mental Health.
Change in self-reported type D (distressed) symptoms using the Type D Scale-14 (TYPE-D), from baseline (Pre) to 6 months follow-up. | Pre (within one month before Intervention week 1), Post (one week after Intervention week 3), 3 month Follow-up, 6 month Follow-up
  The ''distressed'', or Type D, personality combines two basic traits: negative affectivity (NA) and social inhibition (SI). NA refers to individuals with a tendency to experience negative emotions (strongly related to the construct of neuroticism, while SI is the tendency to inhibit emotions and behaviors in social interactions (related to the construct of introversion). The scale consists of seven items each assessing NA and SI (14-items). Participants rate their personality on a 5-point Likert scale by being asked to rate to what degree statements are true for them, on a 5-point scale (0=false; 4=true). A cutoff score of 10 on both the NA and the SI scale is used to classify participants as having a Type D personality.
Change in self-reported suicidal ideation using the Beck Scale for Suicide Ideation (BSI), from baseline (Pre) to 6 months follow-up. | Pre (within one month before Intervention week 1), Post (one week after Intervention week 3), 3 month Follow-up, 6 month Follow-up
  The Beck Scale for Suicide Ideation is a self-report scale comprising 21 items used to detect and measure the intensity of a person's attitudes, behaviors, and plans to commit suicide during the past week. It was developed as a self-report version of the interviewer-administered Scale for Suicide Ideation (SSI). As with the SSI, in the BSI there are five screening items to reduce the need for those not presenting with suicidal ideation from having to complete the entire scale. The ratings for the first 19 items are summed to yield a total score, ranging from 0 to 38.
Change in self-reported interoceptive awareness using the Multidimensional Assessment of Interoceptive Awareness (MAIA), from baseline (Pre) to 6 months follow-up. | Pre (within one month before Intervention week 1), Post (one week after Intervention week 3), 3 month Follow-up, 6 month Follow-up
  Two closely related constructs, body awareness and interoceptive awareness are suggested as potential mediators of the health benefits of mind-body therapies, including, mindfulness meditation, Tai Chi and yoga. This assessment scale comprising 32 items serves to identify and distinguish beneficial and maladaptive body awareness. The MAIA comprises eight subscales: Noticing, Distracting, Worrying, Attention Regulation, Emotional Awareness, Self-Regulation, Body Listening and Trusting.
Change in sustained attention using the Computerized Cognitive Assessment, from baseline (Pre) to 3 months follow-up | Pre (within one month before Intervention week 1), Post (one week after Intervention week 3), 3 month Follow-up
  The participants will perform a sustained attention task in which they identify targets (such as the letter 'x') presented in a series of sequential non-targets (such as the digits 1- 9) either in the center or to either side of a fixation point. During this task, the probe will ask participants to describe their thoughts at intermittent intervals.
Change in diurnal salivary cortisol levels, from baseline (Pre) to 3 months follow-up | Pre (within one month before Intervention week 1), Post (one week after Intervention week 3), 3 month Follow-up
  Cortisol is considered an essential player in understanding stress and stress related effects in the field of psychoneuroendocrinology. Participants will be trained in the routine collection of saliva samples using Salivettes (Sarstedt, Inc, Germany). Participants will be required to collect 8 saliva samples at specified times over the course of 48 hours at Pre, Post, 3 month follow-up.
Change in diurnal salivary α-amylase levels, from baseline (Pre) to 3 months follow-up | Pre (within one month before Intervention week 1), Post (one week after Intervention week 3), 3 month Follow-up
  α-amylase is considered a proxy measure of norepinephrine and epinephrine neurotransmitters involved in the stress response. Thus, α-amylase provides some indication of an individuals level of arousal related to stress. Participants will be trained in the routine collection of saliva samples using Salivettes (Sarstedt, Inc, Germany). Participants will be required to collect 8 saliva samples at specified times over the course of 48 hours at Pre, Post, 3 month follow-up.
Change in salivary cortisol awakening response, from baseline (Pre) to 3 months follow-up | Pre (within one month before Intervention week 1), Post (one week after Intervention week 3), 3 month Follow-up
  Cortisol is considered an essential player in understanding stress and stress related effects in the field of psychoneuroendocrinology. The awakening response indicates an individual's level of arousal at the time of awakening. Participants will be trained in the routine collection of saliva samples using Salivettes (Sarstedt, Inc, Germany). Participants will be required to collect 8 saliva samples at specified times over the course of 48 hours at Pre, Post, 3 month follow-up.
Change in salivary α-amylase awakening response, from baseline (Pre) to 3 months follow-up | Pre (within one month before Intervention week 1), Post (one week after Intervention week 3), 3 month Follow-up
  α-amylase is considered a proxy measure of norepinephrine and epinephrine neurotransmitters involved in reactions to stress. The awakening response indicates an individual's level of arousal at the time of awakening. Participants will be trained in the routine collection of saliva samples using Salivettes (Sarstedt, Inc, Germany). Participants will be required to collect 8 saliva samples at specified times over the course of 48 hours at Pre, Post, 3 month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Yoshio Nakamura, Ph.D., Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Pain Research Center, Salt Lake City, Utah
  - VA Salt Lake City Heath Care System, Salt Lake City, Utah